CLINICAL TRIAL: NCT05760950
Title: China Cohort of Patients With Intracranial Hemorrhage
Brief Title: A Cohort Study of Patients With Intracranial Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Other Study IDs: Cohort Study for ICH
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Routine clinical treatment — Routine clinical treatment is based on the latest international guidelines for intracerebral hemorrhage.

SUMMARY:
As one of the most serious forms of acute stroke, the early mortality rate of intracerebral hemorrhage(ICH) can be as high as 30-40%. The incidence of intracerebral hemorrhage increases with the increase of age. Under the circumstance of the aggravation of aging in China, intracerebral hemorrhage brings a certain burden to families and society.

The results of several studies in recent years have failed to provide new therapeutic approaches for the treatment of cerebral hemorrhage. Therefore, novel therapeutic approaches is urgently needed for ICH. Primary and secondary prevention, acute inpatient care, and poststroke rehabilitation are all critical. The objective of this cohort study is to explore factors that might influence the long-term prognosis of patients with ICH and to further identify new potential targets for intervention.

DETAILED DESCRIPTION:
The observational cohort study will be used to find the possible treatment methods and predictors of functional outcome. The medical records of patients will be collected, including age, sex, comorbid conditions, toxic habits, use of medications (antiplatelets, anticoagulants, and antihypertensives), systolic and diastolic blood pressure, Glasgow Coma Scale (GCS) score, and National Institutes of Health Stroke Scale (NIHSS) score on admission. Image data will also be collected. Follow-up information will be obtained from the medical records or telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Primary intracerebral hemorrhage
* Over 18 year-old

Exclusion Criteria:

* Secondary intracerebral hemorrhage, such as aneurysmal, hemorrhagic transformation of ischemic stroke, cavernomas, arterio-venous malformations, central venous thrombosis, trauma-related, or tumor.
* Pregnant patients.
* Any condition which, in the judgment of the investigator, might increase the risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spontaneous intracerebral hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 90-day
  evaluated by modified Rankin Scale

SECONDARY OUTCOMES:
Neurological deterioration | 14-day
  evaluated by NIHSS or GCS
Functional outcome | 1-year
  evaluated by modified Rankin Scale
Cerebrovascular disease event | 2-year
  ischemic and hemorrhagic events

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, Principal Investigator — Study Principal Investigator Xuanwu Hospital, Beijing
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jolink WM, Klijn CJ, Brouwers PJ, Kappelle LJ, Vaartjes I. Time trends in incidence, case fatality, and mortality of intracerebral hemorrhage. Neurology. 2015 Oct 13;85(15):1318-24. doi: 10.1212/WNL.0000000000002015. Epub 2015 Sep 16. PMID 26377254
- [Result] Greenberg SM, Ziai WC, Cordonnier C, Dowlatshahi D, Francis B, Goldstein JN, Hemphill JC 3rd, Johnson R, Keigher KM, Mack WJ, Mocco J, Newton EJ, Ruff IM, Sansing LH, Schulman S, Selim MH, Sheth KN, Sprigg N, Sunnerhagen KS; American Heart Association/American Stroke Association. 2022 Guideline for the Management of Patients With Spontaneous Intracerebral Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2022 Jul;53(7):e282-e361. doi: 10.1161/STR.0000000000000407. Epub 2022 May 17. No abstract available. PMID 35579034